CLINICAL TRIAL: NCT05014191
Title: Impact of Treatment Positioning on Radiation Therapy RTOG Toxicity in Patients With Vulvar Cancer
Brief Title: Treatment Positioning in Vulvar Cancer Radiation Therapy
Status: Completed | Type: Observational
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 20 KHCC 1111
Record Dates: First submitted 2021-08-14; First posted 2021-08-20 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Radiation therapy in frog leg position
- Radiation therapy in straight leg position

SUMMARY:
The study investigators will conduct a prospective study on patients with non-metastatic vulvar cancer who will receive radiation treatment using Volumetric Arc Therapy (VMAT) modality with curative intent. Our aim is to compare straight-leg versus frog-leg position in terms of RTOG acute skin toxicity. Also, the study investigators will evaluate if positioning has an impact on the total treatment time and deviation on Cone Beam CT (CBCT) that might warrant re-simulation and consequently re-planning.

DETAILED DESCRIPTION:
Vulvar cancer is a rare tumor with a prevalence of about 3-5% of gynecological malignancies with squamous cell carcinoma being the most common histopathologic subtype. It is more common among elderly and postmenopausal women.

Surgery is the cornerstone for the management of patients with early stage vulvar cancer. Radiotherapy is an integral part of the management of vulvar cancer both in the definitive and adjuvant settings.

Several studies have shown that intensity modulated radiotherapy IMRT is associated with better locoregional control compared with 3-dimensional conformal radiotherapy 3DCRT. In addition, it is associated with dosimetric advantage and better sparing of the organs at risk.

Historically, frog-leg position was the standard to provide better access for electron boost in conventional era. After evolution of inverse planning, electron boost is not further needed. Some centers have adopted straight-leg position.

There is paucity of literature regarding vulvar cancer in general and there is lack of data addressing radiation therapy treatment position specifically.

The study investigators will conduct a prospective study on patients with non-metastatic vulvar cancer who will receive radiation treatment using Volumetric Arc Therapy (VMAT) modality with curative intent. Our aim is to compare straight-leg versus frog-leg position in terms of RTOG acute skin toxicity. Also, the investigators will evaluate if positioning has an impact on the total treatment time and deviation on Cone Beam CT (CBCT) that might warrant re-simulation and consequently re-planning.

If both positions proved to be similar in terms of skin toxicity, then the investigators will adopt supine position in the treatment of all patients with vulvar cancer. It will be more comfortable position, and so more reproducible and this reproducibility will be reflected on better treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* ECOG PS = 0-1
* Women with Bx confirmed vulvar cancer FIGO stage I-IVA (treated with curative intent)

Exclusion Criteria:

* Patients whom radiotherapy plans do not cover inguinal lymph nodes will be excluded.

Vulnerable patients will be excluded (pregnant)

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Study Population: Women who were diagnosed with vulvar carcinoma, receiving adjuvant or definitive chemoradiation to primary disease and inguinal lymph nodes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
RTOG acute Skin toxicity (<3 months of starting RT) | 3 months after completion

SECONDARY OUTCOMES:
Total treatment time and the need for re-planning | 3 months for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Fawzi J Abuhijla, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Amman Governorate, Jordan